CLINICAL TRIAL: NCT05299788
Title: The Effectiveness of Active External Warming of Patient Concurrently With Ice Application on the Incision Site on Post-thoracotomy Pain and Analgesic Consumption
Brief Title: Post-thoracotomy Pain Management With Active External Warming and Ice Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Emine Kol, Associated Professor, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 70904504/07
Record Dates: First submitted 2022-02-08; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Post Operative Pain; Pain, Acute; Thoracic Injury
Keywords: Postthoracotomy pain control; Active external warming; Pain management; Ice application; Nursing care
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Thoracic Injuries; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The routine analgesia group (No Intervention): The routine analgesia and warming protocol was applied to patients in the control group.The routine postoperative analgesic treatment protocol at the unit comprises the administration of 75 mg IM (Intramuscular) Diclofenac Sodium before the patient wakes up, 30 mg intravenous (IV) Tramadol if the patient complains of pain when awake (maximum dose of 100 mg/day), and 10 mg/day Morphine Sulfate. In addition to, methods used routinely in the Intensive Care Unit (ICU) such as cotton blankets and socks were used for warming.
- The routine analgesia+active external warming+ice application group (Experimental): In addition to the routine analgesia protocol, the study group was administered non-pharmacological pain control interventions.
  Interventions: Other: Active external warming; Other: Ice application

INTERVENTIONS:
Other: Active external warming — In this study, methods used routinely in the Intensive Care Unit (ICU) such as cotton blankets and socks were used for the control group. In addition to the cotton blankets and socks, electric blankets were used for the patients in the intervention group. In accordance with the literature, the temperature of the electric blanket was set at 38 °C (Celsius) at the beginning and increased to a maximum of 40-41 °C based on the patient's body temperature .
  Arms: The routine analgesia+active external warming+ice application group
Other: Ice application — In the intervention group, an ice pack was applied to the incision site for pain control in addition to active external warming. Ice packs at 0-5 °C with external dimensions of 160 × 91 × 34 mm and a filled weight of 363 g that were kept in the fridge were used for ice application. To prevent direct contact of the ice pack with the patient's skin, the ice pack was wrapped in a thin cotton sheath.
  Arms: The routine analgesia+active external warming+ice application group

SUMMARY:
The aim of study is to investigate the effects of active external warming of patient concurrently with application of ice to incision site on thoracotomy pain and analgesic consumption. The research is a quasi-experimental design with control and study groups.

DETAILED DESCRIPTION:
The study was initiated after obtaining the written approval of the study centers. The center of the study and the hospital where the research was conducted. Written permission was obtained from the hospital management. Within the scope of the research, the research was explained to the participants and their consent was obtained.

The routine analgesia protocol was applied to patients in the control group. In addition to the routine analgesia protocol, the study group was administered non-pharmacological pain control interventions comprising active external warming and ice application. In the Intensive Care Unit (ICU), all patients stayed in the same area without a separator so they could easily observe each other's interventions and hear the conversations occurring during medical intervention. For this reason, the control group was evaluated first. After the last patient in the control group was transferred to the clinic, the study group was evaluated.

Active External Warming: In the literature, the use of electric blankets and warm blowing devices were recommended as the best methods for postoperative active external warming.In this study, methods used routinely in the Intensive Care Unit (ICU) such as cotton blankets and socks were used for the control group. In addition to the cotton blankets and socks, electric blankets were used for the patients in the intervention group. In accordance with the literature, the temperature of the electric blanket was set at 38 °C (Celsius) at the beginning and increased to a maximum of 40-41 °C based on the patient's body temperature.

Application of ice to the incision site: Studies have reported that the cooling effect of ice packs is higher than that of cooled gel packs. In the intervention group, an ice pack was applied to the incision site for pain control in addition to active external warming. Ice packs at 0-5 °C with external dimensions of 160 × 91 × 34 mm and a filled weight of 363 g that were kept in the fridge were used for ice application. In this study, ice packs were applied in the first 12 postoperative hours for 20 minutes every 2 hours, and a parallel pain assessment was performed.

Measurements of body temperature, analgesic consumption, and pain level were made to evaluate the effectiveness of active external warming and ice application. The measurements and follow-up of the patients in the study and control groups in the ICU were carried out by these investigators.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years who were not underweight or obese (body mass index 19-30 kg/m2)
* Patients woke up within the first two postoperative hours, and had been extubated were included in the study group.

Exclusion Criteria:

* Patients in whom hemodynamic stabilization was not achieved 2 hours after thoracotomy,
* patients with Raynaud's phenomenon, neuropathy, or peripheric vascular disease,
* patients who underwent postoperative procedures that directly affect pain levels, such as decortication and thoracic wall resection,
* patients who received preemptive analgesia for pain control,
* patients who received analgesia through pleural, thoracal, and other catheter methods were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Pain score | Pain scoring was initiated when the patient was extubated and until the postoperative 48th hour were recorded
  McGill Pain Questionnaire Short-Form was used for pain assessment. The Verbal Pain Scale, contained in the McGill Pain Questionnaire Short-Form, measured pain intensity at the four-hour mark rating pain of 0 - 5 with 0 = no pain, 1 = mild pain, 2 = discomforting pain, 3 distressing pain, 4 = horrible pain and 5 = excruciating pain.
Analgesic consumption (mg) | Analgesic consumption was started to be recorded when the patient was admitted to the intensive care unit, and until the postoperative 48th hour were recorded
  Algesic consumption: The analgesic consumption of the patient was evaluated with the analgesics used until the postoperative 48th hour. The amount of analgesic administered to the patient was recorded in milligrams.
Body temperature degree | The patient's body temperature was measured in the first four hours postoperatively
  The patient's body temperature was recorded in degrees Celsius.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Kol, Dr, Study Chair — Researher
Locations (1):
- Akdeniz University Hospital, Antalya, Mediterrian, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Information will be shared by Akdeniz University Scientific Research Unit
Supporting Information: CSR
Time Frame: After complated to study
Access Criteria: Information will be shared by Akdeniz University Scientific Research Unit
URL: http://www.akdeniz.edu.tr/